CLINICAL TRIAL: NCT03494426
Title: Radiofrequency Thoracic Sympathectomy for Chronic Postmastectomy Pain; Randomized Placebo Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madona M.NOMAN, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: thoracic sympathectomy
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-07

CONDITIONS: Post-Mastectomy Chronic Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): patients will receive Radiofrequency thoracic sympathectomy then will receive pregabalin ,tramadol,and tricyclic antidepressants
  Interventions: Procedure: radiofrequency thoracic sympathectomy; Drug: pregabalin ,tramadol,and tricyclic antidepressants
- control group (Active Comparator): patients will receive pregabalin ,tramadol,and tricyclic antidepressants
  Interventions: Drug: pregabalin ,tramadol,and tricyclic antidepressants

INTERVENTIONS:
Procedure: radiofrequency thoracic sympathectomy — Under fluoroscopic guidance thoracic sympathectomy will be done as follow
  1. antroposterior view of upper thoracic vertebrae ,cephalo-caudal adjustment of C - arm until aliment of endplates of T2 and T3
  2. oblique view 20 degree under tunnel view RF 10cm 20G 1mm active tip needle is introduced intimately related to vertebral margin
  3. the depth of the needle will be determined under lateral fluoroscopic view the needle is advanced step by step hugging the lateral vertebra l margin until the tip of the needle situated at the middle of the vertebral body . RF lesion 2min 80c will be done and needle is rotated 90 degree on both sides and another two lesions will be done at the end of the procedure 2ml of lidocaine and 20mg of triamcinolone will be injected at each level Post procedure analgesic protocol consisted of either increase or decrease, according to intensity of pain by 50 mg pregabalin and 50 mg tramadole and 25 mg tryptazole, individualized for each patient.
  Arms: interventional group
Drug: pregabalin ,tramadol,and tricyclic antidepressants — patient will receive anti neuropathic medications

SUMMARY:
Postmastectomy pain syndrome (PMPS) is a neuropathic pain that can follow surgical treatment for breast cancer, The antineuropathic medications (antidepressants and anticonvulsants) are disappointing and have low success rate. Continues Radiofrequency lesioning has been reported as treatment for several chronic pain conditions.The concept that the clinical effect of RF was caused by formation of heat had not been challenged. Thermocoagulation of nerve fibers would interfere with the conduction of nociceptive stimuli and pain would be relived. Thoracic sympathectomy has been done for many painful conditions that includes complex regional pain syndrome .It offers the benefit over stellate ganglion block as it blocks the Kuntz fibers that connect to the brachial plexus roots without passing through stellate ganglion.

DETAILED DESCRIPTION:
Postmastectomy pain syndrome (PMPS) is a neuropathic pain that can follow surgical treatment for breast cancer including radical mastectomy, modified radical mastectomy,and segmental mastectomy (lumpectomy) . The pain is distributed in the anterior chest, axilla, and medial and posterior parts of the arm . This pain can be sufficiently severe enough to interfere with sleep and performance of daily activities.

Patients may develop an immobilized arm, which can lead to severe lymph edema, frozen shoulder syndrome, and complex regional pain syndrome. PMPS can result from surgical damage to the intercostobrachial nerve( the lateral cutaneous branch of the second intercostal nerve) that is often resected at mastectomy .

The etiology of persistent pain after mastectomy is unclear, although it is likely multifactorial and may be partially neuropathic in nature . Previous reports of PMPS have suggested a limited number of potential risk factors, which are inconsistent among studies . While surgical factors, including more extensive surgery (mastectomy), axillary lymphnode dissection, and reconstruction have been postulated as important risk factors for chronic pain, many studies do not support this association. Adjuvant treatment, such as radiation, chemotherapy, and hormonal therapy, has also been occasionally associated with persistent pain .

Among demographic factors, younger age correlates with increased incidence of persistent pain in some studies but not others .

The antineuropathic medications (antidepressants and anticonvulsants) are disappointing and have low success rate, also have multiple drawbacks , specifically excessive sedation that affects daily life activities of those patients .

Radiofrequency has been used for interruption of the sympathetic chain to treat intractable pain in the sacral pelvic region or for management of visceral pain and on complex regional pain syndrome.

Radiofrequency has the advantage over surgical resection , in that it is more selective and may cause fewer complications.

Thoracic sympathectomy has been done for many painful conditions that includes complex regional pain syndrome , neuropathic pain of upper limb and it has been done for vasospastic diseases such as Raynaud's phenomenon it offers the benefit over stellate ganglion block as it blocks the Kuntz fibers that connect to the brachial plexus roots without passing through stellate ganglion .

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic post-mastectomy pain for at least 6 month post-operative
* Patients with VAS ≥ 5
* Patients on pregabalin dose ≥ 150 mg daily
* Patients treated with more than one line of anti-neuropathic drugs [e.g. pregabalin+(tricyclic antidepressants or selective serotonin reuptake inhibitors ) or pregabalin+ tramadole]
* Lymphedema of the upper limb

Exclusion Criteria:

* Patient refusal
* Coagulopathy
* Chest and back deformity hindering procedure impossible
* Infection at the introduction site of the needle

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The intensity of pain | up to 3 months after the procedure
  The intensity of pain measured by visual analogue score

SECONDARY OUTCOMES:
The changes in analgesics consumption | 1 month, 2 month and 3 month post-procedure
  The changes in analgesics consumption
The changes in mid-arm circumference | 1 month post- procedure
  The changes in mid-arm circumference
The changes in post-menopausal hot flashes if it was a pre-procedure complaint | 3 month post- procedure
  The changes in post-menopausal hot flashes if it was a pre-procedure complaint

CONTACTS AND LOCATIONS:
Overall Officials: Essam E Abd El Hakem, MD, Study Director — Assiut University; Ashraf A Mohamed, MD, Study Director — Assiut University; Diab F Hetta, MD, Study Director — Assiut University
Locations (1):
- Madona Misheal Boshra Noman, Asyut, Egypt

REFERENCES:
- [Background] Smith WC, Bourne D, Squair J, Phillips DO, Chambers WA. A retrospective cohort study of post mastectomy pain syndrome. Pain. 1999 Oct;83(1):91-5. doi: 10.1016/s0304-3959(99)00076-7. PMID 10506676
- [Background] H. Hoseinzade, A. Mahmoodpoor, D. Agamohammadi, and S. Sanaie, "Comparing the effect of stellate ganglion block and gabapentin on the post mastectomy pain syndrome," Rawal Medical Journal, vol. 33, no. 1, pp. 21-24, 2008.
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Steegers MA, Wolters B, Evers AW, Strobbe L, Wilder-Smith OH. Effect of axillary lymph node dissection on prevalence and intensity of chronic and phantom pain after breast cancer surgery. J Pain. 2008 Sep;9(9):813-22. doi: 10.1016/j.jpain.2008.04.001. Epub 2008 Jun 30. PMID 18585963
- [Background] Carpenter JS, Andrykowski MA, Sloan P, Cunningham L, Cordova MJ, Studts JL, McGrath PC, Sloan D, Kenady DE. Postmastectomy/postlumpectomy pain in breast cancer survivors. J Clin Epidemiol. 1998 Dec;51(12):1285-92. doi: 10.1016/s0895-4356(98)00121-8. PMID 10086821
- [Background] Cohen SP, Sireci A, Wu CL, Larkin TM, Williams KA, Hurley RW. Pulsed radiofrequency of the dorsal root ganglia is superior to pharmacotherapy or pulsed radiofrequency of the intercostal nerves in the treatment of chronic postsurgical thoracic pain. Pain Physician. 2006 Jul;9(3):227-35. PMID 16886031
- [Background] Cahana A, Van Zundert J, Macrea L, van Kleef M, Sluijter M. Pulsed radiofrequency: current clinical and biological literature available. Pain Med. 2006 Sep-Oct;7(5):411-23. doi: 10.1111/j.1526-4637.2006.00148.x. PMID 17014600
- [Background] Guo L, Kubat NJ, Nelson TR, Isenberg RA. Meta-analysis of clinical efficacy of pulsed radio frequency energy treatment. Ann Surg. 2012 Mar;255(3):457-67. doi: 10.1097/SLA.0b013e3182447b5d. PMID 22301609